CLINICAL TRIAL: NCT02752165
Title: Telemedicine Enhanced Asthma Management Through the Emergency Department
Acronym: TEAM-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jill Halterman, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60286
Record Dates: First submitted 2016-03-11; First posted 2016-04-26 (Estimated); Results first posted 2024-02-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- TEAM-ED Intervention Group (Experimental): Facilitation of preventive asthma management through telemedicine assessment and follow-ups in addition to guideline-based provider prompting
  Interventions: Other: TEAM-ED
- Enhanced Usual Care (Active Comparator): Report of symptoms to primary care physician
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: TEAM-ED — Facilitation of preventive asthma management through telemedicine assessment and follow-ups in addition to guideline-based provider prompting
  Arms: TEAM-ED Intervention Group
Other: Enhanced Usual Care — Report of symptoms to primary care physician
  Arms: Enhanced Usual Care

SUMMARY:
In the US, children from minority ethnic and racial backgrounds suffer disproportionately from asthma and account for substantially more emergency department (ED) visits and hospitalizations than non-minority children. While NHLBI guidelines recommend daily preventive medications for all children with persistent asthma to prevent morbidity as well as ED visits and hospitalizations, many children who should receive preventive medications are not receiving them. This is in part because children presenting to the ED for an acute asthma exacerbation rarely receive preventive asthma care, due to the ED's focus on acute, episodic care. The NHLBI guidelines recommend that children follow-up with a primary care provider (PCP) within 1-4 weeks of the ED visit. The post-ED follow-up visit is an opportunity for the PCP to prescribe effective preventive asthma medications, step-up medication for children who demonstrate poor control, promote adherence, and provide education on asthma self-management and trigger control. However, rates for follow-up after an asthma-related ED visit are extremely low, and preventive care is delivered inconsistently even when children are seen in follow-up. In the investigators' prior work they have found that a provider prompting intervention can enhance the delivery of guideline-based preventive asthma treatments at the time of a primary care office visit and ultimately reduce morbidity. They have also found that telemedicine can link children with persistent asthma to a provider for optimal chronic illness management. The goal of this project is to use a novel telemedicine-based program to facilitate primary care follow-up and promote the delivery of guideline-based preventive care for high-risk children presenting to the ED for an asthma exacerbation. The investigators will utilize a 2-group randomized trial to test the TEAM-ED intervention. The intervention includes: 1) a telemedicine assessment at the child's school within one week of discharge from the ED and completed by a PCP, 2) 'point-of-care' prompting to promote the provision of guideline-based preventive care during the telemedicine visit, and 3) two additional telemedicine-assisted follow-up assessments to assure optimal response to treatment and tailor the care regimen as needed. The investigators will assess the effectiveness of the program in reducing respiratory morbidity and improving preventive asthma care, with follow-up assessments at 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Prior physician diagnosis of asthma
* current emergency visit for an acute asthma exacerbation, requiring nebulized albuterol therapy
* Persistent or poor control of asthma, defined by NHLBI guidelines

Exclusion Criteria:

* Inability to speak and understand either English or Spanish
* No access to a phone for follow-up surveys
* Participation in another asthma study at the time of enrollment, or a sibling participating in this or another study Other significant medical conditions that could interfere with assessment of asthma-related measures
* children in foster care or other situations in which consent cannot be obtained from a legal guardian

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JIll Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Halterman JS, Fagnano M, Tremblay P, Butz A, Perry TT, Wang H. Effect of the Telemedicine Enhanced Asthma Management Through the Emergency Department (TEAM-ED) Program on Asthma Morbidity: A Randomized Controlled Trial. J Pediatr. 2024 Mar;266:113867. doi: 10.1016/j.jpeds.2023.113867. Epub 2023 Dec 6. PMID 38065280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in two emergency departments in Rochester, NY in 2016-2021.
Pre-assignment Details: Participants were screened for inclusion/exclusion criteria (age, zip code, asthma severity, reason for emergency visit, foster care, etc.) at the time of the visit to the emergency room. Children were excluded if they did not meet enrollment criteria.
Period: Overall Study
Arm/Group | TEAM-ED Intervention Group | Enhanced Usual Care
Started | 191 | 193
Completed | 146 | 144
Not Completed | 45 | 49
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Protocol Violation | 6 | 5
Not completed — Lost to Follow-up | 33 | 38

BASELINE CHARACTERISTICS:
Population: 10 participants were excluded from analysis as we later learned they did not meet the eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | TEAM-ED Intervention Group | Enhanced Usual Care | Total
Number analyzed (Participants) | 185 | 188 | 373
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (2.6) | 6.5 (1.8) | 6.4 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 75 | 149
  Male | 111 | 113 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 57 | 121
  Not Hispanic or Latino | 121 | 131 | 252
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 94 | 106 | 200
  White | 17 | 15 | 32
  More than one race | 30 | 32 | 62
  Unknown or Not Reported | 40 | 33 | 73
Region of Enrollment [Number; unit: participants]
  United States | 185 | 188 | 373
Mean Symptom-Free Days in prior 2 weeks [Mean (Standard Deviation); unit: days] | 6.61 (4.9) | 6.88 (4.6) | 6.7 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptom-Free Days in the Prior 2 Weeks
Description: Number of days without symptoms in the prior 2 weeks
Time Frame: At the 3-month follow-up assessment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEAM-ED Intervention Group | Enhanced Usual Care
Number analyzed (Participants) | 165 | 157
days | 9.5 (4.9) | 10.1 (4.6)

2. Primary Outcome: Number of Symptom-Free Days in the Prior 2 Weeks
Description: Number of days without symptoms in the prior 2 weeks
Time Frame: At the 6-month follow-up assessment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEAM-ED Intervention Group | Enhanced Usual Care
Number analyzed (Participants) | 161 | 159
days | 10.2 (4.6) | 10.4 (4.3)

3. Primary Outcome: Number of Symptom-Free Days in the Prior 2 Weeks
Description: Number of days without symptoms in the prior 2 weeks
Time Frame: At the 9-month follow-up assessment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEAM-ED Intervention Group | Enhanced Usual Care
Number analyzed (Participants) | 155 | 145
days | 10.4 (4.6) | 10.5 (4.3)

4. Primary Outcome: Number of Symptom-Free Days in the Prior 2 Weeks
Description: Number of days without symptoms in the prior 2 weeks
Time Frame: At the 12-month follow-up assessment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEAM-ED Intervention Group | Enhanced Usual Care
Number analyzed (Participants) | 146 | 144
days | 10.3 (4.8) | 10.0 (4.7)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TEAM-ED Intervention Group | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/189
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/189
Other Adverse Events (participants affected / at risk) | 0/185 | 0/189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT02752165/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT02752165/ICF_001.pdf